CLINICAL TRIAL: NCT05559762
Title: Impact of Regular Night Shift Work on 24-hour Blood Glucose Levels in Nurses
Brief Title: Impact of Night Shift Work on 24-hour Blood Glucose Levels
Status: Completed | Type: Observational
Sponsor: Lincoln Memorial University (Other)
Collaborators: Providence St Joseph Health (Unknown)
Responsible Party: Principal Investigator, Lindsey Miller, Associate Professor, Lincoln Memorial University
Other Study IDs: STUDY2022000529
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Circadian Rhythm; Inversion; Metabolic Disease
MeSH Terms: conditions — Metabolic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Day Shift: Nurses regularly working 12hr day shifts
- Night Shift: Nurses regularly working night shift

SUMMARY:
This study will determine whether nurses regularly working night shifts have elevated 24-hour glucose levels compared to nurses regularly working day shifts, using continuous glucose monitoring (CGM).

ELIGIBILITY:
Inclusion Criteria:

* • RNs working at least a 0.6 FTE and 12-hour night or day shift (not able to alternate between days and nights) for at least the past two months

  * Free from presence of uncontrolled chronic illness and specifically prediabetes, Type 1 or Type 2 diabetes (but not including history of gestational diabetes) and not currently taking any glucose-lowering or steroid medication
  * Not currently pregnant or breastfeeding
  * English speaking and able to provide informed consent
  * Must own and know how to operate a Smartphone
  * Must be willing and able to wear two small sensors attached by adhesive for the study duration, the Fibion SENS activity monitor and the Dexcom G6 continuous glucose monitor
  * Must regularly consume food during shifts and refrain from actively attempting weight loss during the study duration
  * Must work only one job at the time of study participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Full time nurses working either day shifts or night shifts
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
24hr glucose | 7 days
  continuous glucose monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Miller, Principal Investigator — Lincoln Memorial University
Locations (1):
- Providence Sacred Heart Hospital, Spokane, Washington, United States

IPD SHARING:
Plan to Share IPD: No